CLINICAL TRIAL: NCT04948931
Title: The Effect of Aromatherapy Application on Cognitive Functions, Anxiety and Sleep Quality in Elderly People With Diabetes
Brief Title: The Effect of Aromatherapy on Cognitive Functions, Anxiety and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Satı Can, Principal Investigator, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AIBU-SBF-SC-02
Record Dates: First submitted 2021-06-23; First posted 2021-07-02 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; aromatherapy; elderly; anxiety; cognitive function; sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Three groups: Lavender aromatherapy group, rosemary aromatherapy group and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lavender aromatherapy (Experimental): As an intervention to this group, lavender application will be made by inhalation. Participants will apply lavender oil in half an hour before going to bed every night for a month under the supervision of a relative. The application will be done by dripping three drops on cotton, holding it 5-10 cm away from the nose for five minutes and breathing normally.
  Interventions: Other: Lavender aromatherapy
- Rosemary aromatherapy (Experimental): As an intervention to this group, rosemary application will be made by inhalation. Participants will apply rosemary oil in half an hour before going to bed every night for a month under the supervision of a relative. The application will be done by dripping three drops on cotton, holding it 5-10 cm away from the nose for five minutes and breathing normally.
  Interventions: Other: Rosemary aromatherapy
- Control (Placebo Comparator): Distilled water will be used for the application to this group. The application will be made every night for a month, half an hour before going to bed, under the supervision of a relative. Participants will apply distilled water by dropping three drops on cotton, holding it 5-10 cm away from the nose, for five minutes and breathing normally.
  Interventions: Other: Control

INTERVENTIONS:
Other: Lavender aromatherapy — The application will be once a day, every day for four weeks. Each session will take five minutes.
  Arms: Lavender aromatherapy
Other: Rosemary aromatherapy — The application will be once a day, every day for four weeks. Each session will take five minutes.
  Arms: Rosemary aromatherapy
Other: Control — The application will be once a day, every day for four weeks. Each session will take five minutes.
  Arms: Control

SUMMARY:
The aim of this study is to determine the effect of aromatherapy application on cognitive functions, anxiety and sleep quality in elderly people with diabetes.

DETAILED DESCRIPTION:
In addition to its physiological complications, diabetes is a disease that has negative effects on cognitive functions and is accompanied by anxiety and sleep problems. These problems negatively affect diabetes management and glycemic control. Ensuring glycemic control is the most important goal of diabetes treatment. The chronic and progressive nature of diabetes, the continuous increase in the number of individuals with diabetes and the accompanying problems lead the individual to seek alternative treatment methods in addition to clinical medical treatment. When the literature is examined, it is seen that aromatherapy is used in many clinical applications. Studies have shown the positive effects of lavender and rosemary and aromatherapy on cognitive functions, anxiety and sleep problems. However, no comprehensive studies on its effects in the elderly with diabetes were found. This study was planned to determine the effect of aromatherapy application on cognitive functions, anxiety and sleep quality in elderly people with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Who agreed to participate in the research
* Those aged 65 and over
* Diagnosed with diabetes for at least 1 year
* Having no problems with hearing, speaking, seeing and smelling in a way that hinders communication
* Those who have no problem in verbal communication
* Passing the sense of smell test
* Not taking current anxiolytic or hypnotic therapy
* Not diagnosed with a psychiatric illness and without a diagnosis of mental disability
* Do not have any respiratory system disease such as asthma, COPD and allergic skin disease
* No diagnosis of epilepsy disease
* No known allergy to essential oils to be used in the application
* Those who did not use any of the other complementary and integrative application methods at the time of the study.
* Not using sleeping pills

Exclusion Criteria:

* Failure to make interventions within the specified time
* Not attending one of the sessions
* Unwillingness to cooperate with the study
* In addition to existing diseases, respiratory system diseases such as asthma, COPD and allergic diseases
* Known allergy to essential oils and oil used in the study.
* Failed to pass the sense of smell test.
* Receiving anxiolytic or hypnotic therapy
* Those with a diagnosis of psychiatric illness
* Those with a diagnosis of epilepsy disease
* Speech, hearing and vision loss
* Those who do not agree to participate in the research
* Living alone

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Blessed Orientation Memory Concentration Test (BOMCT) | four weeks
  The scale consists of 6 items. It is a test that evaluates the cognitive functions of orientation, memory and concentration. To reach a total score of 28 (worst score) in the scale, the number of errors in the scale in each item is multiplied by the weighted coefficients determined. In the scale evaluation, a point is given to each error in the answers given by the individual, and the total score is obtained by multiplying the scores given differently by the weight points determined differently for each question. An increase in the score indicates a decline in cognitive functions.
Pittsburg Sleep Quality Scale (PUKI) | four weeks
  The scale includes a total of 24 questions and 19 questions are self-report questions and are answered by the individual. Five questions are answered by the spouse or roommate and are not included in the scoring. The 18 items participating in the scoring were grouped into seven components. Each component is evaluated between 0-3 points (0: good, 3: bad). The total score ranges from 0 to 21 and consists of the sum of all components. A high total scale score indicates poor sleep quality. If the total score is 5 or more, it is classified as poor sleep quality, if the total score is between 0-4, the sleep quality is good, and between 5-21, the sleep quality is poor.
Spielberger State-Trait Anxiety Scale (STAI) | four weeks
  The scale consists of two parts:
  1. State Anxiety Scale: It is a 4-point Likert-type scale consisting of 20 questions aiming to measure how individuals feel themselves at the moment. The scores obtained from the scale range from 20 to 80, with high scores indicating high anxiety and low scores indicating low anxiety levels. 0-19 points from the scale indicate that there is no anxiety, 20-39 points indicate mild, 40-59 points moderate, 60-79 points indicate the level of severe anxiety, and a score above 60 indicates the need for professional help.
  2. Trait Anxiety Scale: It indicates how the person feels during the process, regardless of the situation and conditions. The scores obtained from the scale vary between 20 and 80, and a high score indicates a high level of anxiety, and a low score indicates a low level of anxiety. 0-30 indicates low anxiety, 31-49 indicates moderate anxiety, and 50 and higher indicates high anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin YILDIRIM USTA, Prof, Study Director — Bolu Abant Izzet Baysal University, Health Sciences Faculty, Department of Nursing
Locations (1):
- SATI CAN, Bolu, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No